CLINICAL TRIAL: NCT02514850
Title: A Randomised, Single Dose, Double-blind, Double-dummy, Three-period Cross-over Trial to Compare the Pharmacodynamic and Pharmacokinetic Properties of Biochaperone® Combo With Humalog® Mix25 and With Simultaneous Injections of Humalog® and Lantus® in Subjects With Type 2 Diabetes
Brief Title: A Trial to Compare the Pharmacodynamic and Pharmacokinetic Properties of Biochaperone® Combo With Humalog® Mix25 and With Simultaneous Injections of Humalog® and Lantus® in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BC3-CT018
Record Dates: First submitted 2015-07-29; First posted 2015-08-04 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin lispro, isophane insulin lispro drug combination (25:75); Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biochaperone Combo (Experimental): single subcutaneous injection of 0.8 U/kg + injection of placebo (0.9% NaCl) to ensure the double dummy
  Interventions: Drug: Biochaperone Combo; Drug: Placebo
- Humalog Mix25 (Active Comparator): single subcutaneous dose of 0.8 U/kg + injection of placebo (0.9% NaCl) to ensure the double dummy
  Interventions: Drug: Humalog Mix25; Drug: Placebo
- Humalog and Lantus (Active Comparator): simultaneous subcutaneous injections of 0.2 U/kg Humalog and 0.6 U/kg Lantus
  Interventions: Drug: Humalog; Drug: Lantus

INTERVENTIONS:
Drug: Biochaperone Combo — Injection of BioChaperone Combo
  Arms: Biochaperone Combo
Drug: Humalog Mix25 — Injection of Humalog Mix25
  Arms: Humalog Mix25
Drug: Humalog — Injection of Humalog
  Arms: Humalog and Lantus
Drug: Lantus — Injection of Lantus
  Arms: Humalog and Lantus
Drug: Placebo — Injection of saline 0.9% solution
  Arms: Biochaperone Combo; Humalog Mix25

SUMMARY:
This is a single centre, randomised, double-blind, double-dummy, 3-treatment, 3-period cross-over, euglycaemic clamp study in subjects with type 2 diabetes on stable insulin treatment. Each subject will be randomly allocated to a treatment sequence and will be administered single subcutaneous doses of 0.8 U/kg Biochaperone® Combo, 0.8 U/kg Humalog® Mix25 or simultaneous subcutaneous injections of 0.2 U/kg Humalog® and 0.6 U/kg Lantus® during three separate dosing visits.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (as diagnosed clinically) for ≥ 12 months
* HbA1c levels ≤ 9.0%
* Total insulin dose of < 1.2 U/kg/day
* Body mass index between 20.0 and 35.0 kg/m2 (both inclusive)
* Body weight ≤ 125.0 kg
* Fasting serum C-peptide ≤ 1 nmol/L
* Treated with a stable insulin regimen for ≥ 3 months prior to screening

Exclusion Criteria:

* Type 1 diabetes mellitus
* Known or suspected allergy to the trial products or related products
* Previous participation in this trial. Participation is defined as randomised
* Participation in any clinical trial within 3 months prior to this trial
* Clinically significant abnormal haematology, biochemistry, lipids, or urinalysis screening tests, as judged by the Investigator considering the underlying disease
* Supine blood pressure at screening outside the range of 90-160 mmHg for systolic or 50-95 mmHg for diastolic and/or resting supine heart rate outside the range 50 -90 beats per minute. This exclusion criterion also pertains to subjects being on antihypertensives
* Use of GLP-1 receptor agonists or oral antidiabetic drugs (OADs) other than stable intake of metformin within 4 weeks prior to screening
* Women of child bearing potential, not willing to use contraceptive methods

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve (AUCGIR) 12-30h (mg/kg) | from 12h to 30 hours
  Area under the glucose infusion rate curve from 12 hours to 30 hours

SECONDARY OUTCOMES:
AUCGIR 0-last (mg/kg) | Up to 30 hours
  Area under the glucose infusion rate curve from 0 hours until the end of clamp
GIRmax (mg/kg/min) | Up to 30 hours
  Maximum glucose infusion rate
tGIRmax | Up to 30 hours
  Time to maximum glucose infusion rate
AUCLis 0-30h | Up to 30 hours
  Area under the insulin lispro plasma concentration time curve
AUCGla 0-30h | Up to 30 hours
  Area under the insulin glargine plasma concentration time curve
tmax Gla | Up to 30 hours
  Time to maximum insulin glargine plasma concentration
tmax Lis | Up to 30 hours
  Time to maximum insulin lispro plasma concentration
Adverse events | Up to 9 weeks
  Number of adverse events
Hypoglycaemic episodes | Up to 9 weeks
  Number of Hypoglycaemic episodes
Local tolerability | Up to 9 weeks
  Number and intensity of injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, MD, Principal Investigator — Profil Institut Für Stoffwechselfforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany